CLINICAL TRIAL: NCT06645158
Title: Self-Monitoring of Transcutaneous Bilirubinometry in Healthy Term and Near-Term Neonates: a Multi-center Prospective Study
Brief Title: TCB Self-Monitoring in Healthy Term and Near-Term Neonates
Status: Completed | Type: Observational
Sponsor: Neonatal-Infant Brain and Behavior Development Network (Network)
Collaborators: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Multi-TCB
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; transcutaneous bilirubin; neonate
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- normal neonate: gestational age >= 35wk; did not admitted to hospital for any reason; did not need phototherapy within 60h after birth;
  Interventions: Device: Transcutaneous bilirubin level monitoring

INTERVENTIONS:
Device: Transcutaneous bilirubin level monitoring — self-monitoring by parents long-term: from birth to 30 days of age

SUMMARY:
The goal of this observational study is to monitor the transcutaneous bilirubin (TCB) level in healthy near-term and full-term neonates from birth to 30 days of age across China. The main question it aims to answer is:

Development of TcB Nomogram to Identify Neonatal Hyperbilirubinemia in Term and Late-preterm Infants Compare the changing trend of TCB among different areas in China Compare the changing trend of TCB among different gestational groups in China

ELIGIBILITY:
Inclusion Criteria:

Gestational age >=35wk; did not admitted to hospital for any reason Less than 30 days of age

Exclusion Criteria:

Accept phototherapy within 60h of age

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy neonates from participating hospitals from 26 provinces in China
Sampling Method: Probability Sample
Enrollment: 220950 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Development of TcB Nomogram in Term and Late-preterm Infants from birth to 30 days of age | through study completion, an average of 1 year
  From birth to 7 days of age, newborns should undergo transcutaneous bilirubin monitoring twice daily. From 8 to 14 days of age, jaundice should be monitored once daily, and from 14 to 30 days of age, monitoring should be done at least once every two days.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's Medical Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided